CLINICAL TRIAL: NCT03781258
Title: Safety and Feasibility of Transition to Anti-thrombotic Monotherapy With the HeartMate 3 LVAS: A Multicenter Prospective Controlled Study
Brief Title: Anti-thrombotic Monotherapy in HeartMate 3 Left Ventricular Assist System (LVAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Prof. Ivan Netuka, MD, Ph.D., Chairman of the Department of Cardiovascular Surgery, Institute for Clinical and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Version 1.0
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Cardiovascular Diseases
Keywords: Mechanical circulatory support; Anti-thrombotic monotherapy
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — Warfarin

STUDY DESIGN:
Intervention Model Description: Patients implanted with the HeartMate 3 LVAS will be screened for participation in the study with established stability at 6 months after implantation of the device. If inclusion criteria are met, patients will be transitioned to a single anti-thrombotic therapy with Acetylsalicylic Acid (ASA) or equivalent and anticoagulation with warfarin will be withdrawn. ASA will be administered in a minimum dose of 100 mg per day with dosage adjustments based on VerifyNow testing up to a maximum of 200 mg daily. The primary endpoint will be analyzed at 90 and 180 days after initiation of the single antiplatelet therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anit-thrombotic monotherapy (Other): Patients with HeartMate 3 LVAS transitioning from Warfarin and Acetylsalicylic Acid (ASA) therapy to receive anti-thrombotic monotherapy (ASA).
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Anti-thrombotic monotherapy (ASA)-Warfarin withdrawal.

SUMMARY:
The purpose of this prospective controlled study is to obtain a multi-center safety and feasibility data on patients managed with anti-thrombotic monotherapy with HeartMate 3 LVAS.

DETAILED DESCRIPTION:
Patients implanted with the HeartMate 3 LVAS will be screened for participation in the study with established stability at 6 months after implantation of the device. If inclusion criteria are met, patients will be transitioned to a single anti-thrombotic therapy with Acetylsalicylic Acid (ASA) or equivalent antiplatelet therapy and anticoagulation with warfarin will be withdrawn. ASA will be administered in a minimum dose of 100 mg per day with dosage adjustments based on VerifyNow testing up to a maximum of 200 mg daily. The primary endpoints will be analyzed at 90 and 180 days after initiation of the single antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients implanted with HeartMate 3 LVAS irrespective of intended goal of treatment of bridge to transplant or destination therapy
* a minimum of 6 months since HeartMate3 LVAS implantation free of thromboembolic events and pump malfunction
* evidence of forward flow across the aortic valve (with aortic valve opening of at least 1:2 per cardiac cycle) at baseline echocardiography (ECHO) or after speed reduction as long as no evidence of progression of heart failure is noted, based on a combination of biomarkers and clinical assessment follow-up (see Appendix III); Clinical assessment will include review of the biomarkers, invasive or non-invasive hemodynamics (as available or indicated) and clinical physical examination

Exclusion Criteria:

* absence of an informed consent
* presence of any prosthetic valve or central aortic valve repair (e.g. Park's stitch)
* presence of any other ancillary circulatory assist device system
* known history of major thrombotic event e.g. deep vein thrombosis (DVT)
* known history of stroke
* left atrial appendage in patients with atrial fibrillation or flutter not addressed by resection or exclusion at a time of the implant
* evidence of any intracardiac thrombus evidenced by transoesophageal echocardiography
* any other clinical indication for a use of long-term anticoagulation using a vitamin K antagonist or thrombin inhibitor (e.g. specified known genetic thrombotic mutation mandating the therapy, malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival free of a pump malfunction due to thrombosis or any ischemic stroke | 180 days
  To determine survival free of a pump malfunction due to thrombosis or any ischemic stroke at 90-days (primary safety end point) and at 180-days (primary efficacy end point) in patients implanted with HeartMate 3 LVAS after transition to a single antithrombotic with Acetylsalicylic Acid (ASA) or equivalent antiplatelet therapy.

SECONDARY OUTCOMES:
Adverse Events | 180 days
  Adverse events rates per Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) definitions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague 4, Czechia

REFERENCES:
- [Background] Mehra MR, Goldstein DJ, Uriel N, Cleveland JC Jr, Yuzefpolskaya M, Salerno C, Walsh MN, Milano CA, Patel CB, Ewald GA, Itoh A, Dean D, Krishnamoorthy A, Cotts WG, Tatooles AJ, Jorde UP, Bruckner BA, Estep JD, Jeevanandam V, Sayer G, Horstmanshof D, Long JW, Gulati S, Skipper ER, O'Connell JB, Heatley G, Sood P, Naka Y; MOMENTUM 3 Investigators. Two-Year Outcomes with a Magnetically Levitated Cardiac Pump in Heart Failure. N Engl J Med. 2018 Apr 12;378(15):1386-1395. doi: 10.1056/NEJMoa1800866. Epub 2018 Mar 11. PMID 29526139
- [Background] Netuka I, Ivak P, Tucanova Z, Gregor S, Szarszoi O, Sood P, Crandall D, Rimsans J, Connors JM, Mehra MR. Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the MAGENTUM 1 study. J Heart Lung Transplant. 2018 May;37(5):579-586. doi: 10.1016/j.healun.2018.03.002. Epub 2018 Apr 11. PMID 29655662
- See also: Two-Year Outcomes with a Magnetically Levitated Cardiac Pump in Heart Failure — http://www.nejm.org/doi/pdf/10.1056/NEJMoa1800866
- See also: Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the Minimal AnticoaGulation EvaluatioN To aUgment heMocompatibility (MAGENTUM) 1 study — http://doi.org/10.1016/j.healun.2018.03.002